CLINICAL TRIAL: NCT03427047
Title: A Prospective, Randomized Study Comparing Surgical and Economic Parameters of Total Knee Replacement Performed Using Two Different Surgical Techniques: Medacta MyKnee® Surgical Technique Using Efficiency Single-use Instruments Versus Stryker Navigation Surgical Technique Performed With Conventional Metal Instruments.
Brief Title: Comparing Surgical and Economical Parameters of Total Knee Replacement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyKnee 20170612
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Osteo Arthritis Knee; Total Knee Arthroplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MyKnee with single use Efficiency Instrument (Active Comparator): Patients randomized in this group will undergo Total Knee Arthroplasty utilizing patient matched cutting blocks and single use instruments. Customization will be by a CT scan of patients knee.
  Interventions: Device: MyKnee with single use Efficiency Instrument
- Stryker Navigational with conventional metal instruments (Active Comparator): Patients randomized in this group will undergo Total Knee Arthroplasty with conventional metal instruments. CT scan are not utilized with this arm.
  Interventions: Device: Stryker Navigational with conventional metal instruments

INTERVENTIONS:
Device: MyKnee with single use Efficiency Instrument — Total Knee Arthroplasty utilizing a CT scan for customization of cutting blocks with single use instrumentation
  Arms: MyKnee with single use Efficiency Instrument
Device: Stryker Navigational with conventional metal instruments — Total Knee Arthroplasty without customization of cutting blocks using conventional metal instruments.
  Arms: Stryker Navigational with conventional metal instruments

SUMMARY:
Randomized study comparing surgical and economic parameter of Total Knee Arthroplasty performed using two different specific surgical techniques.

DETAILED DESCRIPTION:
Randomized 1: ratio study comparing Medacta MyKnee surgical technique using Efficiency single use instruments versus Stryker Navigation surgical techniques performed with conventional instruments. MyKnee surgical technique patients will receive a CT scan of the surgical knee which enables custom manufacturing of the MyKnee cutting blocks. Stryker Navigational surgical technique patients will not require a CT scan. Both groups of patients will undergo total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years 2) BMI ≤35 3) Undergoing unilateral total knee arthroplasty due to osteoarthritis (primary or post-traumatic OA) with the Medacta GMK Sphere 4) Able and willing to give consent and to comply with study requirements, including follow up visit at 6 weeks

Exclusion Criteria:

* Is participating in another clinical study 2) Has inflammatory arthritis 3) Has knee avascular necrosis 4) Has severe deformity, defined as greater than 15 degrees varus or 10 degrees valgus relative to the mechanical axis. 5) Has retained hardware in the knee that requires removal and interferes with TKA procedure 6) Has prior high tibial osteotomy (HTO)

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hur, MD, Principal Investigator — Forte Sports Medicine and Orthopedics
Locations (1):
- Methodist Sports Medicine Research & Education Foundation, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Started | 46 | 36
Completed | 46 | 34
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments | Total
Number analyzed (Participants) | 46 | 36 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 16 | 41
  >=65 years | 21 | 20 | 41
Age, Continuous [Mean (Full Range); unit: years] | 64.32 [53 to 75] | 65.67 [50 to 75] | 64.99 [50 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 16 | 8 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 46 | 36 | 82

OUTCOME MEASURES:

1. Primary Outcome: Compare Time-saving Associated With the Two Procedures.
Description: Measure clean up time at end of surgery in minutes
Time Frame: Day of surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 36
minutes | 25.12 [8.00 to 52.33] | 28.47 [10.00 to 130.10]

2. Primary Outcome: Patient OR Time From Both Study Arms
Description: Measure skin to skin, tourniquet time and femoral and tibial resection time in minutes
Time Frame: Day of surgery
Population: Number analyzed differs due to uncollected data
Measure: Mean (Full Range); unit: minutes
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 36
minutes
  incision to closure time: number analyzed (Participants) | 45 | 35
  incision to closure time | 69.83 [51.47 to 97.32] | 70.44 [58.42 to 82.82]
  tourniquet time | 53.07 [41.98 to 78.48] | 52.84 [27.25 to 92.03]
  femur and tibia time: number analyzed (Participants) | 46 | 7
  femur and tibia time | 10.98 [4.68 to 30.08] | 11.87 [0.83 to 19.80]

3. Secondary Outcome: Estimated Blood Loss From Both Study Arms
Description: Volume of estimated blood loss in cc's
Time Frame: Day of surgery
Measure: Mean (Full Range); unit: cc's
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 36
cc's | 105.43 [50 to 200] | 100 [50 to 200]

4. Secondary Outcome: Baseline of Hemoglobin Both Study Arms
Description: Measure in grams per deciliter
Time Frame: Baseline, 1 day post-op or at discharge from hospital
Measure: Mean (Full Range); unit: grams per deciliter
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 36
grams per deciliter
  Baseline | 14.18 [12.20 to 16.30] | 13.77 [11.40 to 15.70]
  Post-op | 12.57 [10.70 to 15.20] | 12.31 [9.60 to 15.60]

5. Secondary Outcome: Volume of Transfusions Both Study Arms
Description: Measure amount of blood patient receives in ML
Time Frame: Day of surgery
Measure: Mean (Full Range); unit: mL
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 36
mL | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Instrument Trays Sent to Sterilization Both Study Arms
Description: Record number of trays sent to be sterilized
Time Frame: Day of surgery
Measure: Mean (Full Range); unit: trays
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 36
trays | 5.48 [3 to 7] | 9.5 [7 to 20]

7. Secondary Outcome: Amount of Waste From Surgery Both Study Arms
Description: Combined weight of recyclable and non-recyclable waste in grams
Time Frame: Day of surgery
Measure: Mean (Full Range); unit: grams
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 36
grams | 20196.7 [14242.8 to 27442.3] | 17653.5 [13108.8 to 20910.6]

8. Secondary Outcome: Baseline of Mechanical Axis Both Study Arms
Description: Determine radiographic analysis by measuring knee mechanical axis in degrees
Time Frame: Baseline, post-operative 6 weeks
Population: Data only available for 44 of 46 participants in Myknee arm
Measure: Mean (Full Range); unit: degrees
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 44 | 34
degrees
  Baseline | 6.05 [0 to 12] | 5.71 [0 to 15]
  Post-operative 6 weeks | 1.64 [0 to 6] | 1.24 [0 to 7]

9. Secondary Outcome: Change From Baseline of Tibial Slope Both Study Arms
Description: Determine radiographic analysis by measuring tibial angles in degrees
Time Frame: Baseline, post-operative 6 weeks
Measure: Mean (Full Range); unit: degrees
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 44 | 34
degrees
  Baseline | 3.80 [0 to 12] | 2.08 [0 to 8]
  Post-operative 6 weeks | 1.8 [0 to 8] | 1.87 [0 to 4]

10. Secondary Outcome: Related Complications
Description: Assess adverse events and serious adverse events related to both procedures
Time Frame: Baseline, day of surgery, post-op 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
Number analyzed (Participants) | 46 | 34
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks post-op
Arm/Group | MyKnee With Single Use Efficiency Instrument | Stryker Navigational With Conventional Metal Instruments
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/36
Other Adverse Events (participants affected / at risk) | 3/46 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MyKnee With Single Use Efficiency Instrument (N=46) | Stryker Navigational With Conventional Metal Instruments (N=36)
Acute posterior knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Weepy Left Knee Incision (Surgical and medical procedures) | 0 (0) | 1 (1)
Extremely stiff with swelling and pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT03427047/Prot_SAP_000.pdf